CLINICAL TRIAL: NCT03741517
Title: Prospective Longitudinal Observation Trial of Clinical and Molecular Features of Pancreatic Neuroendocrine Tumours
Brief Title: Biomarker Study of Pancreatic Neuroendocrine Tumours
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Joakim Crona, Associate Professor, Uppsala University
Other Study IDs: PRORESS pancreas
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Biopsy, Large-Core Needle; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: 18F-FDG-PET — Fludeoxyglucose F18
Radiation: 68Ga-DOTATOC-PET — DOTA-tyr3-Octreotide Ga68
Radiation: Computed tomography — Computed tomography of thorax and abdomen with 3-phase contrast
Other: Core needle biopsy — Core needle biopsy of metastatic lesions
Other: Phlebotomy — Phlebotomy from peripheral vein

SUMMARY:
The biology of pancreatic neuroendocrine tumors can change during the disease course. This evolution of disease can manifest through increases in tumor proliferation rate, resistance to medical therapy and/or a change in tumor hormone secretion. This study aims to characterize how the biology of pancreatic neuroendocrine tumors change over time, measured by; patient symptoms, biochemistry, contrast enhanced computed tomography, DOTATOC-PET, FDG-PET and core needle biopsy with histopathological analysis (Ki67 index and tumor cell differentiation). Uptake on 68Ga-DOTATOC and 18F-FDG-PET will be correlated directly to tumor cell proliferation rate. Fraction of patients with spatial heterogeneity in DOTATOC as well as FDG uptake as well as metachronous changes in all collected data will be documented. Biomaterial from whole blood and core needle biopsies will be characterized on the molecular level, and those findings will be integrated to the above specified clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed consent
* Pathology confirmed diagnosis of pancreatic neuroendocrine tumor WHO grade 1-3 or neuroendocrine carcinoma grade 3.

Exclusion Criteria:

* Patient does not consent
* Pregnancy or no contraceptive in fertile women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic Neuroendocrine Tumors
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Protocol adherence | Study inclusion
  Defined as the proportion of patients where that following investigations are performed: Core needle biopsy, FDG-PET, DOTATOC-PET, research blood samples, pancreatic hormones and hormonal syndromes.

OTHER OUTCOMES:
Safety of core needle biopsy: NCI Common Terminology Criteria | At study inclusion and within 48 hours of the procedure
  Defined as a NCI Common Terminology Criteria for Adverse Events 4.03 grade 3-4 adverse event related to the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska Sjukhuset, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes